CLINICAL TRIAL: NCT02700022
Title: A Phase I/Ib Study of Alisertib Plus R-EPOCH for Treatment of Myc-Positive Aggressive B-Cell Lymphomas
Brief Title: A Phase I Study of Alisertib + R-EPOCH for Treatment of Myc-Positive Aggressive B-cell Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1503
Record Dates: First submitted 2016-02-17; First posted 2016-03-07 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicular Lymphoma; Burkitt Lymphoma
Keywords: Lineberger Comprehensive Cancer Center; Alisertib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Burkitt Lymphoma | interventions — MLN 8237; Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alisertib combined with R-EPOCH (Experimental): Dose escalation will take place within cohorts. Subjects will receive alisertib tablets twice daily in combination with R-EPOCH chemotherapy on days 1 through 5 of each 21-day cycle. The treatment will be given in 6 cycles. The first 3 patients to be enrolled will receive a 20 milligram (mg) dose of alisertib. The dose of alisertib will be increased or decreased as more subjects enter the study. Each dose level will be evaluated for safety and tolerability before the next higher dose is given. The dose levels will be modified until the maximum tolerated dose (MTD) is reached. Once the MTD has been established, enrollment into that cohort will continue with up to a maximum of 24 patients total enrolled into the study.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Dose escalation of alisertib: level 1 - 20 mg, level 2 - 30 mg, level 3 - 40 mg PO BID on Days 1-5 of six 21-day cycles, combined with R-EPOCH Rituximab, IV infusion on day 1 of each cycle; Etoposide, IV infusion for 96 hours on days 1, 2, 3, and 4 Doxorubicin, IV infusion for 96 hours on days 1, 2, 3, and 4 Vincristine, IV infusion for 96 hours on days 1, 2, 3, and 4 Cyclophosphamide, IV infusion for 15 minutes on day 5 Prednisone, PO daily on days 1, 2, 3, 4, and 5
  Other Names: Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone

SUMMARY:
This phase I/Ib study is designed to establish the safety and maximum tolerated dose (MTD, which will also be the recommended phase II dose (RP2D)) of the aurora kinase A inhibitor alisertib when combined with dose-adjusted (DA)-R-EPOCH (rituximab, etoposide, doxorubicin, vincristine, cyclophosphamide and prednisone) in patients with CD20-positive diffuse large B-cell lymphoma (DLBCL), transformed follicular lymphoma or Burkitt lymphoma positive for Myc gene rearrangement (Myc+). Filgrastim or peg-filgrastim is also included with each cycle of R-EPOCH. Once we identify the MTD, an expansion cohort limited to the Myc+ DLBCL population will be opened to further characterize clinical activity and safety.

Secondary objectives include estimates of complete response rate (CR) and progression free survival (PFS). We will also explore for associations between baseline kinome signatures and/or RNA sequencing and CR, and identify differential kinome and transcriptome prior to and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 y/o (no upper age limit)
* ECOG PS ≤2
* Disease - Histologically or cytologically documented newly diagnosed (stages II, III or IV) Myc-positive DLBCL, transformed follicular lymphoma, or high-grade unclassifiable with features intermediate between DLBCL and Burkitt lymphoma
* Myc Positive lymphoma is defined by:

  * Positive for Myc gene rearrangement by fluorescence in-situ hybridization (FISH) involving various breakpoints (e.g. 8-14, 8-22 and 2-8) AND concurrent gene rearrangements in bcl-2 and/or bcl-6 by FISH OR
  * Myc and Bcl-2 overexpression defined by > 40% Myc and > 70% Bcl-2 expression by IHC. Patients may enroll in the study based on the local laboratory evaluation, but these should be confirmed by the UNC Hematopathology Laboratory retrospectively
* Positive for CD20 via immunophenotyping
* Prior Treatment: Previously untreated or who received a maximum of one cycle of combination chemotherapy (i.e. R-CHOP, R-EPOCH, or R-hyperCVAD) within 4 weeks of study entry except patients who require dose reduction after the first cycle of off-study R-EPOCH.
* Measurable disease as assessed by 2 dimensional measurements by CT (≥ 1.5 cm).
* Adequate organ function as demonstrated by:

  * Bone marrow function (without platelet transfusion or myeloid growth factor support within two weeks of screening) as demonstrated by:
  * Hemoglobin ≥ 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelet count ≥75,000/mm3
* And hepatic and renal function as demonstrated by:

  * Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN); ALT and AST up to 5 x ULN if liver metastases present
  * Total serum bilirubin ≤1.5 x ULN
  * Serum creatinine ≤1.5 x ULN or CrCl of ≥ 30
* Adequate renal function as defined by: Calculated creatinine clearance must be ≥ 30 mL/minute based on Cockcroft-Gault formula
* Documented negative serologic testing for human immunodeficiency virus (HIV), hepatitis B (unless serologically positive due to prior vaccination), and hepatitis C within the year prior to enrollment (note: for guidance in defining active infection for hepatitis B, please refer to the WHO guidelines. (World Health Organization, Global Alert and Response (GAR), Hepatitis B (who.int/csr/disease/hepatitis/ whocdscsrlyo20022/en/index4.html)
* Patient agrees to consume no more than 1 standard unit of alcohol per day during the study and for 30 days from the last dose of alisertib. A standard unit of alcohol is defined as a 12 oz beer (350 mL), 1.5 oz (45 mL) of 80-proof alcohol, or one 6-oz (175 mL) glass of wine.
* Women of childbearing potential (WOCBP) must have negative pregnancy test within 7 days prior to D1 of treatment
* Female subjects must be:

  * Post-menopausal for at least one year before the screening visit, or
  * Surgically sterilized, or
  * Willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject, even if surgically sterilized (ie, status post-vasectomy), agrees to:

  * Use an acceptable method for contraception (effective barrier contraception or:
  * Completely abstain from heterosexual intercourse) during the entire study treatment period through 4 months after the last dose of alisertib.
* Ability to swallow oral medications
* As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study
* Sufficient data to calculate the International Prognostic Index (IPI) score at baseline:

  * Age
  * Stage of Disease
  * LDH
  * ECOG performance status
  * number of extranodal sites
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Adequate left ventricular function with ejection fraction ≥ 40% by echocardiogram or MUGA scan.

Exclusion Criteria

* CNS involvement of DLBCL
* Major surgery within 4 weeks prior to entry
* Receiving any other concurrent cytotoxic, biologic agent(s) or investigational agent ; NOTE: Concurrent intrathecal chemotherapy for CNS prophylaxis allowed per institutional standards
* Receipt of investigational drugs within 14 days before D1 of alisertib
* Prior administration of an Aurora A kinase-targeted agent, including alisertib
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers, non-invasive bladder cancer, "low risk" adenocarcinoma of the prostate and carcinoma in situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib and during the study.
* Radiation therapy to more than 25% of the bone marrow (note: whole pelvic radiation is considered to be over 25%)
* Prior allogeneic bone marrow or organ transplantation
* Known GI disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib; examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen
* Requirement for constant administration of proton pump inhibitor from 5 days prior to D1 of alisertib, and/or requirement for constant administration of H2 antagonist, or pancreatic enzymes; intermittent uses of antacids or H2 antagonists are allowed
* Requirement for drugs, juices and/or herbs strongly inhibit CYP3A4 from within 7 days prior to D1 of alisertib and throughout treatment NOTE: Glucocorticoids are considered inducers of CYP3A4. However, their use is allowed if patient has been taking a continuous dose of no more than 15 mg/day of prednisone (or its equivalent) for at least 1 month prior to D1 of alisertib. In addition, low dose steroid use for the control of nausea and vomiting will be allowed. Topical steroid use and inhaled steroids are also permitted.
* Systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Female subject who is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening (within 7 days prior to D1 of treatment). Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
* Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to alisertib.
* Administration of myeloid growth factors or platelet transfusion within 14 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years

SECONDARY OUTCOMES:
Toxicity | from day 1 of treatment until up to 2 years after treatment
  Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0
Rate of Response | from day 1 of treatment until up to 2 years after treatment
  Rate of CR will be evaluated as defined by The International Harmonization Project for Response Criteria
Progression free survival | from day 1 of treatment until up to 2 years after treatment or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dittus, DO, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hills, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/